CLINICAL TRIAL: NCT06448611
Title: Identification and Characterization of Circulating Tumor Cells Before and After Treatment in a Cohort of Patients Treated for Resectable Stage I-III Merkel Cell Carcinoma
Brief Title: Identification and Characterization of Circulating Tumor Cells Before and After Treatment (Surgery and Radiotherapy) in a Cohort of Patients Treated for Resectable Stage I-III Merkel Cell Carcinoma
Acronym: MERCCALIBI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL23_0452
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Merkel Cell Carcinoma
Keywords: Circulating Tumor Cells
MeSH Terms: conditions — Carcinoma, Merkel Cell; Neoplastic Cells, Circulating | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of Patients Treated for Resectable Stage I-III Merkel Cell Carcinoma: Entire cohort
  Interventions: Other: Blood Test

INTERVENTIONS:
Other: Blood Test — Research and quantification of Circulating Tumor Cells

SUMMARY:
The goal of this prospective observational study is to evaluate the presence of circulating tumoral cells in patients over 18 with a stage I-III resectable Merkel cell carcinoma after the initial therapeutic sequence of surgery and radiotherapy. The main question it aims to answer is :

Can any residual disease be found in the form of circulating tumoral cells in blood samples of patients treated with surgery and radiotherapy for a resectable, stage I to III Merkel cell carcinoma ? When possible, the circulating tumoral cells count will be compared to the one realized in a blood sample of the same patient before surgery and radiotherapy.

Participants will :

* Have a blood sample taken before surgery (if the patient is addressed to our center early enough),
* Have a blood sample taken immediately after surgery and radiotherapy (for all).
* Two additional blood samples will be taken during the 6-months and 12-months visit to set up a biobank.

DETAILED DESCRIPTION:
The main goal of this study is to evaluate the presence of circulating tumoral cells in patients circulating tumoral cells after surgery and radiotherapy in patients with stage I to III Merkel cell carcinoma.

Another goal will be to track changes in the number of circulating tumoral cells before and after treatment in patients with stage I to III Merkel cell carcinoma, who have had a blood sample taken before starting treatment.

Investigators will also set up a biobank, which is a collection of blood samples taken every six months for one year. These samples will help with future research.

The study will include patients over 18 years old with stage I to III Merkel cell carcinoma, treated at the Dermatology Departments of Montpellier and Nimes University Hospitals. Investigators will not include pregnant or breastfeeding women, patients not covered by social security, those under court protection, those unable to give consent, or those with stage IV Merkel cell carcinoma or stage I to III Merkel cell carcinoma where complete remission is not possible. All patients will give free and informed consent to participate.

Patients will be divided into two groups based on when they are referred to the university hospital for treatment.

Group A: If the tumor is fully removed before the patient is referred to the hospital.

Group B: If the tumor is still present when referred to the hospital. This can happen if:

* Only a biopsy has been done to confirm the tumor.
* The tumor was removed but it is stage III with lymph node involvement. Both scenarios will not affect the main goal (checking for circulating tumoral cells after treatment). However, the change in circulating tumoral cell numbers before and after treatment can only be checked in Group B, where patients had a blood sample taken before treatment.

Both groups will have follow-up visits at 6 and 12 months. The main endpoint will be the circulating tumoral cell detection rate, which is the presence of circulating tumoral cells in their blood right after surgery and radiotherapy. Another measure will be the change in the number of circulating tumoral cells before and after treatment for those who had a blood sample taken before starting treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old
* Patients managed for stage I to III Merkel cell carcinoma,
* For whom complete remission by complete surgical resection is planned (group B) or has been achieved recently, within 6 weeks prior to the inclusion visit (group A).

Exclusion Criteria:

* Pregnant or breast-feeding women
* Failure to obtain written informed consent after a reflection period
* Participant in another research study with an ongoing exclusion period
* Not affiliated to a social security scheme
* Persons under court protection
* Patients unable to give consent, protected adults, vulnerable persons
* Stage IV disease or stage I to III disease for which complete remission is not envisaged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed for stage I to III Merkel cell carcinoma, for whom complete remission by complete surgical resection is planned (group B) or has been achieved recently, within 6 weeks prior to the inclusion visit (group A).
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Circulating tumoral cells detection rate | 6 weeks or less after the therapeutic sequence of surgery and radiotherapy
  Rate of patients with the presence of at least one CTC detected in the peripheral blood directly after the therapeutic sequence of surgery and radiotherapy, in absolute value

SECONDARY OUTCOMES:
Change in the number of pre- and post-therapeutic circulating tumoral cells | 6 weeks or less after the therapeutic sequence of surgery and radiotherapy
  Difference between the number of post-therapeutic CTCs (after surgery and radiotherapy) and the number of pre-therapeutic CTCs (for patients for whom a pre-therapeutic sample was available: group B patients), in absolute value

IPD SHARING:
Plan to Share IPD: No